CLINICAL TRIAL: NCT06713395
Title: Analysis of the Effects of PERMA-Based Integrated Psychological Intervention on Negative Emotions, Treatment Adherence, and Complications in Postoperative Glioma Patients
Brief Title: PERMA-Based Intervention on Negative Emotions, Adherence, and Complications in Postoperative Glioma Patients
Acronym: Glioma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yang Huang (Other Government)
Collaborators: The Affiliated Brain Hospital of Nanjing Medical University (Other Government)
Responsible Party: Sponsor-Investigator, Yang Huang, The Affiliated Brain Hospital of Nanjing Medical University, The Affiliated Brain Hospital of Nanjing Medical University
Organization: The Affiliated Brain Hospital of Nanjing Medical University (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2020-KY091-01
Record Dates: First submitted 2024-11-22; First posted 2024-12-03 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Glioma
Keywords: PERMA; Glioma; Integrated psychological intervention; SAS; SDS; complication
MeSH Terms: conditions — Glioma

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- control group (Other): The control group was provided with standard postoperative care
  Interventions: Other: The control group received standard postoperative care
- observation group (Other): The observation group received an additional PERMA-based integrated psychological intervention
  Interventions: Other: PERMA

INTERVENTIONS:
Other: The control group received standard postoperative care — standard postoperative care
  Arms: control group
Other: PERMA — 1. Establishment of the Integrated Psychological Intervention Team:
     The team consisted of 2 primary nurses, 4 specialist nurses, 1 psychologist, 2 physicians at the attending level or higher, and 2 researchers.
     Team Responsibilities: The primary and specialist nurses were responsible for implementing the intervention protocol. The physicians handled any adverse reactions experienced by the patients. The researchers were in charge of developing the intervention protocol and collecting data. All team members were required to undergo specialized training from the psychologist and pass an assessment before initiating the intervention.
  2. Protocol Development:
     The intervention protocol, including specific content, team responsibilities, implementation process, and responses to adverse events, was carefully developed in written form by the researchers. The protocol was discussed and approved by all team members before implementation.
  3. Protocol Implementation:
  Emotional Support Intervention:
  Arms: observation group

SUMMARY:
The goal of this clinical trial is to evaluate whether a PERMA-based integrated psychological intervention can reduce negative emotions, enhance treatment adherence, and decrease the risk of complications in postoperative glioma patients.

The main questions it aims to answer are:

Can the PERMA-based psychological intervention significantly improve anxiety and depression scores in postoperative glioma patients? Does the intervention improve treatment adherence, reduce complications, and enhance quality of life compared to standard care? Researchers will compare an observation group receiving the PERMA-based psychological intervention to a control group receiving standard postoperative care to see if the intervention improves patient outcomes.

Participants will:

Receive either standard postoperative care (control group) or PERMA-based psychological intervention for one month (observation group).

Be assessed on:

Self-Rating Depression Scale (SDS) and Self-Rating Anxiety Scale (SAS). Treatment Adherence Scale and Complication Record Form. Quality of Life Scale. Be followed for complications using Kaplan-Meier survival analysis.

ELIGIBILITY:
Inclusion Criteria:

* ①Meeting the relevant diagnostic criteria from the 5th edition of the World Health Organization Classification of Central Nervous System (CNS) Tumors, and confirmed through postoperative pathological examination;
* ②Underwent surgical treatment;
* ③Clear consciousness, with good communication ability, and capable of cooperating with healthcare personnel to complete the study;
* ④Complete clinical data.

Exclusion Criteria:

* ①Concurrent diagnosis of other malignant tumors;
* ②Coexisting cognitive impairment or other psychiatric disorders;
* ③Combined liver or kidney dysfunction, immune system disorders, or other severe diseases;
* ④Presence of infectious diseases;
* ⑤Pregnant or breastfeeding women.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2022-01-10 (Actual); Primary Completion 2024-02-15 (Actual); Study Completion 2024-02-25 (Actual)

PRIMARY OUTCOMES:
SAS score | After the four-week intervention
  Self-rating anxiety scale is a widely used psychological assessment tool designed to evaluate an individual's level of anxiety. There are 20 things on the scale, and a score of 100 is the total, assessing various anxiety-related emotions experienced by the participant over the past week. Each item is rated on a 4-point Likert scale, ranging from "no anxiety" to "extremely severe anxiety," where higher scores indicate more severe anxiety. Prior to and one month following the intervention, the SAS scores for each group were documented.
SDS score | After the four-week intervention
  Self-rating depression scale is a commonly used psychological assessment tool designed to evaluate an individual's level of depression. The scale typically consists of 20 items, with a total score of 100, covering various aspects of depression. Using a 4-point Likert scale that goes from "no depression" to "extremely severe depression," participants describe their moods over the course of the previous week. Higher scores signify more severe depression. The SDS scores for both groups were recorded before and one month after the intervention.
treatment adherence | After the four-week intervention
  Complete adherence: The patient actively cooperated with the medical and nursing staff, followed all prescribed treatments and interventions, and complied with medication, examinations, and other medical recommendations on a daily basis. Partial adherence: The patient generally cooperated with the medical and nursing staff but may not have fully adhered to all instructions. Non-adherence: The patient showed poor cooperation, requiring multiple reminders and explanations to comply with treatment protocols. The adherence rate was calculated as the sum of the complete and partial adherence rates. Adherence was recorded one month after the intervention.
Incidence of postoperative complications | During the four-week intervention
The World Health Organization Quality of Life Brief Scale scores | After the four-week intervention
  WHOQOL-BREF is a tool used to assess an individual's quality of life. This scale consists of 26 items, each with five options, rated from 1 to 5, with higher scores reflecting better outcomes (or from very satisfied to extremely dissatisfied). However, items 3, 4, and 26 are reverse-scored. Additionally, there are separate scores for family friction, appetite, and self-assessed survival quality. The scale covers four domains: physical health, psychological health, social relationships, and environment. Participants rate their experiences over the past two weeks. Each domain score is calculated by summing the relevant item scores and standardizing them, yielding a range from 0 to 100, with higher scores indicating better quality of life.

SECONDARY OUTCOMES:
general characteristics | At the time of patient enrollment
  Index: Gender, Age (years), BMI/ (kg/m2), Degree of education, History of diabetes, History of high blood pressure.

CONTACTS AND LOCATIONS:
Locations (1):
- The Affiliated Brain Hospital of Nanjing Medical University, Nanjing, Jiangsu, China